CLINICAL TRIAL: NCT05990673
Title: Determination of the 50% and 95% Effective Dose of Remimazolam for Intravenous Anesthesia Induction in Pediatric Patients
Brief Title: Dose of Remi in Children
Acronym: DRINK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XJH-A-20230606
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia
Keywords: general anesthesia; anesthesia induction; remimazolam
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- remimazolam (Experimental): remimazolam is given for anesthesia induction
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — remimazolam is given intravenously
  Other Names: remimazolam besylate

SUMMARY:
Remimazolam has demonstrated the potential as a valuable medication for procedural sedation and general anesthesia. However, the effective dosage of remimazolam in pediatric patients is still unknown.

ELIGIBILITY:
Inclusion Criteria:

* age from 3 to 12 years old
* patients scheduled for surgery under general anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists status >=Ⅲ
* Body mass index>=28kg/m2
* patients who cannot cooperate with intravenous anesthesia induction
* patients with risk of difficult airway
* patients who are allergic to benzodiazepines
* patients with delayed neurologic function

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
half effective dosage | from injection of remimazolam to loss of consciousness, at an average of 5 minutes
  the dosage by which half of the patients will be sedated

SECONDARY OUTCOMES:
95% effective dosage | from injection of remimazolam to loss of consciousness, at an average of 5 minutes
  the dosage by which 95% of the patients will be sedated

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tan H, Lou AF, Wu JE, Chen XZ, Qian XW. Determination of the 50% and 95% Effective Dose of Remimazolam Combined with Propofol for Intravenous Sedation During Day-Surgery Hysteroscopy. Drug Des Devel Ther. 2023 Jun 13;17:1753-1761. doi: 10.2147/DDDT.S406514. eCollection 2023. PMID 37333966